CLINICAL TRIAL: NCT01210417
Title: Trauma Heart to Arm Time
Acronym: THAT
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 179_06/2010
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Trauma; Hypovolemia; Hemorrhage
Keywords: Trauma; Hypovolemia; Hemorrhage; Out of hospital trauma
MeSH Terms: conditions — Wounds and Injuries; Hypovolemia; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Trauma victims: All prehospital traumatic patients enrolled by our Helicopter Emergency Medical System (HEMS)
  Interventions: Other: Non invasive monitoring

INTERVENTIONS:
Other: Non invasive monitoring — Three-lead electrocardiogram (ECG), PPG oxymetry, non-invasive blood pressure (NIBP) are registered

SUMMARY:
In the prehospital setting it would be helpful to assess primary changes in central blood volume or preload (venous return, stroke volume, diastolic ventricular volume) that occur during the stability phase following injury when regulatory mechanisms are still functioning.

Obviously in this setting a non invasive bedside beat-to-beat index would be helpful.

Pulse Transit Time (PTT) is the sum of Pre-Ejection Period (PEP), the time interval between the onset of ventricular depolarization and the ventricular ejection, and Vascular Transit Time (VTT), the time it takes for the pulse wave to travel from the aortic valve to the peripheral arteries (Obrist et al. 1979). PEP variations are known to correlate with reductions in central blood volume induced by head-up tilt (Chan et al., 2007b, 2008). The same authors also demonstrated that PTT variations follow closely PEP variations and therefore central blood volume variations (Chan et al., 2007b). Following central blood volume reductions induced by head-up tilting ventricular diastolic filling time increases involving an increase in PEP and PTT. Chan et al. (Chan et al., 2007b) concluded that PTT could have been used to assess early central hypovolemia and suggested that joint analysis of PTT and RR intervals could help in predicting the extent of blood volume loss. The investigators hypothesized that sympathetic drive associated with trauma would act on cardiac contractility through beta activity thus shortening PTT without reducing RR interval to the same extent in healthy hearts. We also hypothesized that progressive hypovolemia would lead to a rising of PTT (augmented diastolic filling time) and a RR interval shortening (relative tachycardia). In this study the investigators propose and index based on the beat-to-beat PTT/RR ratio to assess central hypovolemia in traumatic patients enrolled by our Helicopter Emergency Medical System (HEMS) in a prehospital setting.

ELIGIBILITY:
Inclusion Criteria:

* all trauma victims enrolled by our Helicopter Emergency Medical System (HEMS)

Exclusion Criteria:

* need of immediate life-saving manoeuvres as decided by onboard physician following Prehospital Trauma Care (PTC) criteria (CITATION PTC)
* Cardiac arrest
* presence of preexisting chronic illnesses involving the autonomic nervous system such as hypertension, diabetes and any neurological disease
* any preexisting medical therapy including those administered by the emergency medical team as defined in point 1)
* presence of supraventricular ectopic beats more than 5% of total recorded beats
* absence of sinus rhythm
* presence of intraventricular or bundle branch blocks or artificial pacemaker
* spinal chord trauma above D2
* patient age <18 years
* presence of burns not allowing monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All trauma victims enrolled by our Helicopter Emergency Medical System (HEMS)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-09; Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- A.R.E.U. - A.A.T. 118 Milano, Milan, Italy